CLINICAL TRIAL: NCT01806428
Title: THE Activated Protein C (aPC) TREATMENT IMPROVES MICROCIRCULATION IN SEVERE SEPSIS/ SEPTIC SHOCK SYNDROME
Brief Title: Activated Protein C and Microcirculation
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Collaborators: Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Associate Professor, Università Politecnica delle Marche
Other Study IDs: 208249
Record Dates: First submitted 2013-03-06; First posted 2013-03-07 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Severe Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- aPC treatment group: Septic patients with at least two sepsis-induced organ failures occurring within 48 hours of the onset of sepsis treated with activated protein C at 24 mcg/Kg/h for 96 hours
- Control group: Septic patients with at least two sepsis-induced organ failures occurring within 48 hours of the onset of sepsis not treated with activated protein C because of contraindications

SUMMARY:
Objective: to test the hypothesis that recombinant activated protein C (aPC) therapy improves the microcirculation of severe septic patients.

Design: Prospective, open study. Setting: University 12-beds intensive care unit. Patients: Septic patients with at least two sepsis-induced organ failures occurring within 48 hours of the onset of sepsis were included in a one year period.

Interventions: Patients who had no contraindication to aPC administration received aPC at a dose of 24 mcg/kg/h for 96 hours. Patients with contraindications to aPC infusion were considered as controls.

ELIGIBILITY:
Inclusion Criteria:

* Septic patients with at least two sepsis-induced organ failures occurring within 48 hours of the onset of sepsis

Exclusion Criteria:

* hematologic or advanced malignancies
* liver cirrhosis
* severely impaired consciousness (Glasgow Coma Scale score <7 of 15)
* therapeutic limitations (do-not-resuscitate orders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Septic patients with at least two sepsis-induced organ failures occurring within 48 hours of the onset of sepsis
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Microcirculatory Flow Index (MFI) before during and after aPC infusion | 102 hours
  Microcirculatory Flow Index detected in vivo by side-dark field imaging at sublingual microcirculation. It represents the quality of blood flow at microcirculatory level. This study wants to verify any of the considered different types of blood transfused can improve MFI.

SECONDARY OUTCOMES:
Perfused Vessel Density before during and after aPC infusion | 102 hours
  Perfused Vessel Density (PVD) detected in vivo by side-dark field imaging at sublingual microcirculation. It represents the quantity of well perfused vessels at microcirculatory level. This study wants to verify any of the considered different types of blood transfused can improve PVD.
Tissue oxygen saturation (StO2) upslope before during and after aPC infusion | 102 hours
  StO2 upslope is measured with Near InfraRed Spectroscopy at the tenar muscle. It represents the velocity of the recovery of the tissue oxygen saturation after a short period of ischemia of the hand, the Vascular Occlusion Test.

CONTACTS AND LOCATIONS:
Locations (1):
- University ICU, AOU Ospedali Riuniti Ancona, Torrette Di Ancona, Ancona, Italy

REFERENCES:
- [Result] Donati A, Damiani E, Botticelli L, Adrario E, Lombrano MR, Domizi R, Marini B, Van Teeffelen JW, Carletti P, Girardis M, Pelaia P, Ince C. The aPC treatment improves microcirculation in severe sepsis/septic shock syndrome. BMC Anesthesiol. 2013 Sep 26;13(1):25. doi: 10.1186/1471-2253-13-25. PMID 24070065